CLINICAL TRIAL: NCT01732536
Title: A Clinical Evaluation of the Safety and Efficacy of the Steroid-Releasing S8 Sinus Implant Used in Post-Sinus Surgery Patients With Recurrent Sinus Obstruction
Brief Title: Steroid-Releasing S8 Sinus Implant for Recurrent Nasal Polyps
Acronym: RESOLVE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Intersect ENT (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P500-1012
Record Dates: First submitted 2012-11-14; First posted 2012-11-26 (Estimated); Results first posted 2018-07-20 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Chronic Sinusitis; Nasal Polyps
Keywords: corticosteroid-eluting sinus implant; chronic rhinosinusitis; mometasone furoate; polyposis
MeSH Terms: conditions — Nasal Polyps | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants were blindfolded and earmuffed during the baseline procedure and follow-up endoscopic examinations. Implants were removed at Day 60 to allow blinded assessment of bilateral polyp grade at Day 90 by a centralized videoendoscopy review by a panel of 3 independent sinus surgeons.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- S8 Sinus Implant (Experimental): In-office bilateral placement of the S8 Sinus Implant (mometasone furoate, 1350 mcg) in the ethmoid sinuses
  Mometasone furoate nasal spray (200mcg) once daily
  Interventions: Drug: S8 Sinus Implant; Drug: Mometasone furoate nasal spray
- Control (Sham Comparator): In-office bilateral sham procedure
  Mometasone furoate nasal spray (200mcg) once daily
  Interventions: Procedure: Sham procedure; Drug: Mometasone furoate nasal spray

INTERVENTIONS:
Drug: S8 Sinus Implant — In-office bilateral placement of the S8 Sinus Implant (mometasone furoate, 1350 mcg) in the ethmoid sinuses
  Other Names: SINUVA (mometasone furoate) sinus implant
  Arms: S8 Sinus Implant
Procedure: Sham procedure — In-office bilateral sham procedure
  Arms: Control
Drug: Mometasone furoate nasal spray — Two sprays in each nostril once daily, totaling 200 mcg of mometasone furoate throughout Day 90
  Other Names: Nasonex Nasal Spray

SUMMARY:
The RESOLVE Study is a randomized controlled trial with the S8 Sinus Implant in 100 chronic sinusitis patients with recurrent nasal polyps.

DETAILED DESCRIPTION:
RESOLVE is a randomized (1:1), sham-controlled, parallel group, double-blind multicenter study in 100 chronic sinusitis patients who had prior endoscopic sinus surgery and presented with recurrent nasal polyps. The objective of the study was to assess the safety and efficacy of the S8 Sinus Implant, a steroid-eluting sinus implant, consisting of a bioabsorbable self-expanding sinus implant coated with 1350 mcg of mometasone furoate (MF) and a single-use delivery system. Implant is placed in-office in the ethmoid sinus under local anesthesia. The coating on the S8 implant provides controlled release of MF to the sinus mucosa over 90 days, with the majority of drug released within 60 days.

ELIGIBILITY:
Inclusion Criteria

Candidates for this study had to meet ALL of the following inclusion criteria:

1. General Inclusion Criteria

1. Patient has provided written informed consent using a form approved by the reviewing IRB.
2. Patient is ≥ 18 years of age.
3. Patient is willing and able to comply with protocol requirements.
4. Patient has a previous confirmed diagnosis of CS defined as inflammation of the mucosa of the paranasal sinuses.
5. Patient has undergone bilateral total ethmoidectomy (must be at least 90 day beyond the date of last sinus surgery).
6. Patient has recurrent bilateral sinus obstruction due to polyposis (Grades 1 through 3 only).
7. Patient must have a Grade 2 polyposis on at least 1 ethmoid side.
8. Patient is able to tolerate the use of Nasonex topical intranasal steroid spray once daily.
9. Patient is indicated for a repeat ESS per the study definition. Patient must have: (i) a minimum symptom burden on the SNOT 22, consisting of a minimum score of 2 on at least 2 of the 5 hallmark symptoms of CS (nasal blockage, post-nasal discharge, thick nasal discharge, facial pain/pressure, and decreased sense of smell); (ii) persistent symptoms of CS despite ongoing treatment with topical intranasal steroid irrigations or sprays at least once daily for at least 2 weeks preceding enrollment; (iii) had treatment with a high-dose form of steroids (e.g., oral, parenteral, injection into polyps) and/or sinus steroid irrigations within the preceding 2 years, or refused such therapy due to intolerance/side effects; (iv) a known history of repeated courses of treatment with aggressive steroid therapy for recurrent sinusitis; and (v) endoscopic evidence of polyp recurrence, scarring, and/or obstructive mucosal edema.
10. Patient is able to tolerate use of topical/local anesthesia and the implant procedure in an office or clinic setting.
11. In the opinion of the physician, treatment with S8 Sinus Implant or sham procedure is technically feasible (able to pass 5-9 mm device into middle meatus) bilaterally.
12. Female patients of child-bearing potential must not be pregnant and must agree to not become pregnant during the course of the study.
13. Female patients of child-bearing potential must agree to use consistent and acceptable method/s of birth control during the course of the study.

Exclusion Criteria

Candidates were excluded if they met ANY of the following criteria:

General Exclusion Criteria

1. Patient had bilateral total ethmoidectomy less than 90 days previously.
2. Patient had Propel implanted postoperatively less than 90 days previously.
3. Patient has presence of adhesions/synechiae Grades 3 or 4.
4. Patient has presence of severe scarring or adhesions within the ethmoid cavity itself.
5. Patient has presence of Grade 4 polyposis.
6. Patient has known history of immune deficiency (e.g., IGG] subclass deficiency or IGA deficiency, HIV).
7. Patient has concurrent condition requiring active chemotherapy and/or immunotherapy management for the disease (e.g., cancer, HIV, etc.).
8. Patient has oral-steroid dependent condition such as chronic obstructive pulmonary disease (COPD), asthma or other condition.
9. Patient has known history of allergy or intolerance to corticosteroids or mometasone furoate (MF).
10. Patient has known history of resistance or poor response to oral steroids.
11. Patient has presence of physical obstruction that would preclude access to either ethmoid sinus for device delivery (e.g., severe septal deviation, septal spur, very small middle meatus, total obstruction of the nasal passage with severe scarring, polyposis).
12. Patient has clinical evidence of acute bacterial sinusitis (e.g., acute increase in purulent discharge, fever, facial pain etc.).
13. Patient has clinical evidence or suspicion of invasive fungal sinusitis (e.g., bone erosion on prior CT scan, necrotic sinus tissue, etc.).
14. Patient has evidence of disease or condition expected to compromise survival or ability to complete follow-up assessments during the 6 month follow-up period.
15. Patient is currently participating in or recently participated in another clinical trial (within the last 30 days).
16. Patient has history of insulin dependent diabetes mellitus.
17. Patient has previously undergone ESS and experienced a CSF leak or has residual compromised vision as a result of a complication in a prior ESS procedure.
18. Patient has completely resected middle turbinate.
19. Patient has known dehiscence of the lamina papyracea.
20. Patient has evidence of active viral illness (e.g., tuberculosis, ocular herpes simplex, chickenpox, or measles).

    Ocular Exclusion Criteria
21. Patient has history or diagnosis of glaucoma or ocular hypertension (baseline or a known prior ocular exam indicating IOP >21 mm Hg)
22. Patient has closed angle (with or without the presence of peripheral anterior synechiae on gonioscopy)
23. Patient has presence in either eye of: (i) posterior subcapsular cataract, (ii) nuclear sclerosis of Grade +3 or higher; or (iii) cortical cataract of Grade +3 or higher.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith D Forwith, MD, Principal Investigator — Advanced ENT and Allergy; Joseph K Han, MD, Principal Investigator — Eastern Virginia Medical School Department of Otolaryngology
Locations (19):
- United States (19):
  - California Sinus Centers, Atherton, California
  - Cedars-Sinai Medical Center, Sinus Center of Excellence, Los Angeles, California
  - Sacramento Ear, Nose and Throat, Sacramento, California
  - Colorado Ear, Nose, Throat & Allergy, Colorado Springs, Colorado
  - South Florida ENT Associates, Miami, Florida
  - ENT of Georgia, Atlanta, Georgia
  - Northwestern University, Department of Otolaryngology-Head & Neck Surgery, Chicago, Illinois
  - Advanced ENT & Allergy, Louisville, Kentucky
  - Summit Medical Group, Berkeley Heights, New Jersey
  - Albany ENT & Allergy Services, Albany, New York
  - ENT and Allergy Associates, Lake Success, New York
  - Piedmont Ear, Nose & Throat Associates, Winston-Salem, North Carolina
  - Oregon Health and Science University-Dept. of Otolaryngology Head and Neck Surgery, Portland, Oregon
  - Bethlehem ENT Specialty Physicians Associates, Bethlehem, Pennsylvania
  - University of Pennsylvania, Dept of Otolaryngology-Head & Neck Surgery, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Intermountain Ear, Nose & Throat Center, Salt Lake City, Utah
  - Eastern Virginia Medical School Department of Otolaryngology, Norfolk, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No
No plan

REFERENCES:
- [Background] Han JK, Forwith KD, Smith TL, Kern RC, Brown WJ, Miller SK, Ow RA, Poetker DM, Karanfilov B, Matheny KE, Stambaugh J, Gawlicka AK. RESOLVE: a randomized, controlled, blinded study of bioabsorbable steroid-eluting sinus implants for in-office treatment of recurrent sinonasal polyposis. Int Forum Allergy Rhinol. 2014 Nov;4(11):861-70. doi: 10.1002/alr.21426. Epub 2014 Sep 29. PMID 25266981
- [Result] Forwith KD, Han JK, Stolovitzky JP, Yen DM, Chandra RK, Karanfilov B, Matheny KE, Stambaugh JW, Gawlicka AK. RESOLVE: bioabsorbable steroid-eluting sinus implants for in-office treatment of recurrent sinonasal polyposis after sinus surgery: 6-month outcomes from a randomized, controlled, blinded study. Int Forum Allergy Rhinol. 2016 Jun;6(6):573-81. doi: 10.1002/alr.21741. Epub 2016 Mar 14. PMID 26992115

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between January 2013 and November 2013 at 18 clinical sites (12 private, 6 academic).
Pre-assignment Details: A total of 100 patients were enrolled and randomized. met final eligibility. There was a 2-week run-in period before screening during which participants were required to use an intranasal corticosteroid spray.
Groups:
- Treatment: In-office bilateral placement of the S8 Sinus Implant (mometasone furoate, 1350 mcg) in the ethmoid sinuses
- Control: In-office bilateral sham procedure
Period: Overall Study
Arm/Group | Treatment | Control
Started | 53 | 47
Completed | 52 | 46
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment: In-office bilateral placement of the S8 Sinus Implant (mometasone furoate, 1350 mcg) in the ethmoid sinuses
  Mometasone furoate nasal spray (200mcg) once daily
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 53 | 47 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (12.61) | 51.6 (13.12) | 49.6 (12.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 16 | 40
  Male | 29 | 31 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 49 | 46 | 95
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 2 | 8
  White | 47 | 44 | 91
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 53 | 47 | 100

OUTCOME MEASURES:

1. Primary Outcome: Nasal Obstruction/Congestion Score
Description: Nasal Obstruction by patients using a paper questionnaire on a scale from 0 (no problem) to 5 (problem as bad as it can be). Negative values for change from baseline represented reduction (improvement) in
Time Frame: 90 days
Population: Intent-to-treat population. Values were adjusted for steroid and surgical interventions by LOCF approach. There were 3 (3%) participants (1 treatment, 2 control) with missing values at Day 90. No imputation of missing values was performed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 53 | 47
units on a scale
  Baseline | 3.62 (1.180) | 3.30 (1.159)
  Day 90: number analyzed (Participants) | 52 | 45
  Day 90 | 2.31 (1.422) | 2.62 (1.336)
  Change from baseline: number analyzed (Participants) | 52 | 45
  Change from baseline | -1.33 (1.465) | -0.67 (1.446)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p = 0.1365, ANCOVA; Based on between group comparison using ANCOVA model with baseline as a covariate and site and treatment as fixed effects
Statistical Analysis 2: Comparison: Treatment vs Control; The change from baseline to Day 90 in Nasal Obstruction/Congestion score in the subset of participants with higher polyp burden at baseline (grade 2 or higher polyps on each side; N=67); Test type: Superiority; p = 0.0505, ANCOVA — Based on between group comparison using ANCOVA model with baseline as a covariate and site and treatment as fixed effects

2. Primary Outcome: Bilateral Polyp Grade
Description: Polyp grade was determined by a panel of 3 independent sinus surgeons based on a centralized, blinded videoendoscopy review. Each sinus was graded from 0 (no visible polyps) to 4 (nasal polyps completely obstructing nasal cavity) and then the left and right values were added to obtain a total bilateral polyp grade, ranging from 0 to 8. Negative values for change from baseline represented reduction (improvement) in bilateral polyp grade.
Time Frame: 90 days
Population: Intent-to-treat population. Values were adjusted for steroid and surgical interventions by LOCF approach. There were 2 (2%) participants (2 treatment, 0 control) with missing values. No imputation of missing values was performed. Negative values for change from baseline represent improvement.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 53 | 47
units on a scale
  Baseline: number analyzed (Participants) | 51 | 47
  Baseline | 4.90 (0.918) | 4.39 (1.448)
  Day 90: number analyzed (Participants) | 52 | 47
  Day 90 | 4.12 (1.162) | 4.00 (1.720)
  Change from baseline: number analyzed (Participants) | 51 | 47
  Change from baseline | -0.76 (0.875) | -0.38 (0.998)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p = 0.0985, ANCOVA; Based on ANCOVA model with baseline as a covariate, site and treatment as fixed effect
Statistical Analysis 2: Comparison: Treatment vs Control; Bilateral polyp grade change in a subset of 67 patients with higher polyp burden at baseline (grade 2 or higher on each side confirmed by the independent panel); Test type: Superiority; p = 0.0490, ANOVA; Based on ANCOVA model with baseline as a covariate, site and treatment as fixed effect

3. Secondary Outcome: Ethmoid Sinus Obstruction
Description: Percentage of the ethmoid sinus volume obstructed by scarring, polyps, or edema on endoscopy, as determined by a panel of 3 independent sinus surgeons based on a centralized, blinded videoendoscopy review using a 100-mm visual analogue scale (VAS), ranging from 0 (absence of obstruction) to 100 (complete obstruction). Negative values for change from baseline represented reduction (improvement) in ethmoid sinus obstruction.
Time Frame: 90 days
Population: Intent-to-treat population. Values were adjusted for steroid and surgical interventions by LOCF approach. There was1 (1.0%) participant (treatment) with missing values at baseline and Day 90. No imputation of missing values was performed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | S8 Sinus Implant | Control
Number analyzed (Participants) | 53 | 47
units on a scale
  Baseline: number analyzed (Participants) | 52 | 47
  Baseline | 70.59 (18.201) | 62.74 (25.673)
  Day 90: number analyzed (Participants) | 52 | 47
  Day 90 | 53.54 (20.140) | 57.17 (28.516)
  Change from baseline: number analyzed (Participants) | 52 | 47
  Change from baseline | -17.05 (19.361) | -5.57 (18.279)
Statistical Analysis 1: Comparison: S8 Sinus Implant vs Control; Test type: Superiority; p = 0.0099, ANCOVA

4. Secondary Outcome: Bilateral Polyp Grade
Description: Polyps were graded by clinical investigators on a scale from 0 (no visible polyps) to 4 (nasal polyps completely obstructing nasal cavity) and then the left and right values were added to obtain a total bilateral polyp grade, ranging from 0 to 8. Negative values for change from baseline indicate reduction (improvement) in nasal polyps.
Time Frame: 90 days, 6 months
Population: Intent-to-treat population. Values were adjusted for steroid and surgical interventions by LOCF approach. There were 3 (3.0%) participants (1 treatment, 2 control) with missing values at 90 days and 4 (4.0%) participants (2 treatment, 2 control) with missing values at Month 6. No imputation of missing values was performed.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | S8 Sinus Implant | Control
Number analyzed (Participants) | 53 | 47
units on a scale
  Baseline | 4.68 (0.956) | 4.32 (1.105)
  90 days: number analyzed (Participants) | 52 | 45
  90 days | 3.65 (1.655) | 4.24 (1.667)
  Change from baseline to 90 days | -1.04 (1.680) | -0.09 (1.203)
  Month 6: number analyzed (Participants) | 51 | 45
  Month 6 | 3.96 (1.587) | 4.36 (1.708)
  Change from baseline to 6 months: number analyzed (Participants) | 51 | 45
  Change from baseline to 6 months | -0.71 (1.527) | 0.02 (1.158)
Statistical Analysis 1: Comparison: S8 Sinus Implant vs Control; Test type: Superiority; p = 0.0162, ANCOVA — P-value for change from baseline to 90 days not adjusted for multiplicity; ANCOVA model with baseline as a covariate and site and treatment as fixed effects
Statistical Analysis 2: Comparison: S8 Sinus Implant vs Control; Test type: Superiority; p = 0.0175, ANCOVA — P-value for change from baseline to 6 months not adjusted for multiplicity; ANCOVA model with baseline as a covariate and site and treatment as fixed effects

5. Secondary Outcome: Nasal Obstruction Symptom Evaluation (NOSE) Score
Description: NOSE scale is a validated symptom scoring instrument consisting of 5 questions each scored by patients on a 5-point Likert scale from 0 (not a problem) to 4 (severe problem), then multiplied by 5 and resulting in a total score ranging from 0 to 100. Negative values for change from baseline represented reduction (improvement) in NOSE score.
Time Frame: 6 months
Population: Intent-to-treat population. Values were adjusted for steroid and surgical interventions by LOCF approach. There were 3 (3.0%) participants (1 treatment, 2 control) with missing values at Month 6. No imputation of missing values was performed.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- S8 Sinus Implant: Bilateral in-office placement of the S8 Sinus Implant (mometasone furoate, 1350 mcg) in the ethmoid sinuses and continued Nasonex (mometasone furoate nasal spray, 200 mcg)
  S8 Sinus Implant: Bilateral in-office placement of S8 sinus implant with 1350 mcg of mometasone furoate and continued steroid nasal spray (mometasone furoate, 200 mcg) once daily
- Control: Bilateral in-office sham procedure in the ethmoid sinuses and continued Nasonex (mometasone furoate nasal spray, 200 mcg)
  Sham procedure: Bilateral in-office sham procedure and continued steroid nasal spray (mometasone furoate, 200 mcg) once daily
Arm/Group | S8 Sinus Implant | Control
Number analyzed (Participants) | 53 | 47
units on a scale
  Baseline | 66.79 (26.658) | 63.19 (23.943)
  Month 6: number analyzed (Participants) | 52 | 45
  Month 6 | 41.83 (24.395) | 50.67 (25.597)
  Change from baseline: number analyzed (Participants) | 52 | 45
  Change from baseline | -25.58 (28.174) | -12.22 (23.874)
Statistical Analysis 1: Comparison: S8 Sinus Implant vs Control; Test type: Superiority; p = 0.0209, ANCOVA — P-value not adjusted for multiplicity; Based on between arm comparison using ANCOVA model with baseline as a covariate and site and treatment as fixed effects

6. Secondary Outcome: Percentage of Patients Indicated for Revision Endoscopic Sinus Surgery (RESS)
Description: To be indicated for RESS, the following criteria had to be met:
  * Continued to use topical intranasal steroids daily;
  * Continued to complain of at least 2 symptoms of chronic sinusitis despite ongoing topical intranasal steroid use
  * Needed or had received at least 1 course of aggressive steroid therapy or had refused such therapy due to intolerance/side effects; and
  * Had endoscopic evidence of persisting ethmoid sinus obstruction (bilateral polyp grade >=2 on at least one side)
Time Frame: 90 days, 6 months
Population: Intent-to-treat population consisted of all patients in whom an implant or sham procedure was attempted. There were 2 (2.0%) participants (1 treatment, 1 control) who withdrew from the study prior to Day 90. No imputation of missing values was performed.
Measure: Count of Participants; unit: Participants
Arm/Group | S8 Sinus Implant | Control
Number analyzed (Participants) | 53 | 47
Participants
  Baseline | 53 | 47
  Day 90: number analyzed (Participants) | 52 | 46
  Day 90 | 25 | 36
  Month 6: number analyzed (Participants) | 52 | 46
  Month 6 | 36 | 41

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment though month 6
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/53 | 1/47
Other Adverse Events (participants affected / at risk) | 38/53 | 36/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=53) | Control (N=47)
Suicidal ideation (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=53) | Control (N=47)
Chronic Sinusitits (Infections and infestations) | 11 | 14
Upper respiratory tract infection (Infections and infestations) | 5 | 2
Acute sinusitis (Infections and infestations) | 8 | 11
Nasopharyngitis (Infections and infestations) | 3 | 3
Headache (Nervous system disorders) | 3 | 2
Presyncope (Nervous system disorders) | 2 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 3

LIMITATIONS AND CAVEATS:
1. Absence of defined medical regimen prior to enrollment
2. Investigators grading polyps and assessing indication for RESS were not blinded
3. Indication for RESS at baseline allowed for 1 sinus side to have polyp grade >=1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No